CLINICAL TRIAL: NCT05950802
Title: Optimizing lymphoDepletion to Improve Outcomes In Patients Receiving CAR T Cell Therapy With Yescarta/AxicabtageNeciloleucel (ODIN)
Brief Title: Optimizing lymphoDepletion to Improve Outcomes In Patients Receiving Cell Therapy With Yescarta
Acronym: ODIN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OZM-124
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in two stages: the dose escalation stage to assess the safety and tolerability of a modified LD regimen, and once the MTD is determined, a cohort expansion phase to further characterize the toxicity and efficacy profile and determine the RP2D. The study will enroll approximately 18-24 patients in the dose escalation stage (Part 1), and approximately 20 further patients at cohort expansion (Part 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cyclophosphamide and fludarabine, standard dose (No Intervention): Fludarabine 30mg/m2 Cyclophosphamide 500mg/m2 Days -4, -3, -2
- Cyclophosphamide and fludarabine, standard dose with radiation (Experimental): Fludarabine 30mg/m2 Cyclophosphamide 500mg/m2 Days -6, -5, -4, and 2 Gy in 2 Fractions Days -3, -2
  Interventions: Drug: Cyclophosphamide; Radiation: TLI
- Cyclophosphamide (intermediate dose) and fludarabine (Experimental): Fludarabine 30mg/m2 Cyclophosphamide 750mg/m2 Days -4, -3, -2
  Interventions: Drug: Cyclophosphamide
- Cyclophosphamide (intermediate dose) and fludarabine with radiation (Experimental): Fludarabine 30mg/m2 Cyclophosphamide 750mg/m2 Days -6, -5, -4, and 2 Gy in 2 Fractions Days -3, -2
  Interventions: Drug: Cyclophosphamide; Radiation: TLI

INTERVENTIONS:
Drug: Cyclophosphamide — Higher dose than traditional conditioning chemo
  Other Names: cytoxin, neosar
  Arms: Cyclophosphamide (intermediate dose) and fludarabine; Cyclophosphamide (intermediate dose) and fludarabine with radiation; Cyclophosphamide and fludarabine, standard dose with radiation
Radiation: TLI — radiation given with conditioning chemo
  Arms: Cyclophosphamide (intermediate dose) and fludarabine with radiation; Cyclophosphamide and fludarabine, standard dose with radiation

SUMMARY:
This is a Phase 1b study of participants with Diffuse Large B Cell Lymphoma (DLBCL). The purpose of this study is to identify an optimized lymphodenpletion (LD) regimen by evaluating standard and intermediate doses of Fludarabine (Flu) / Cyclophosphamide (Cy) with or without a fixed dose of total lymphoid irradiation (TLI) in the setting of standard of care CAR T cell therapy.

DETAILED DESCRIPTION:
Patients will be enrolled in two stages: the dose escalation stage to assess the safety and tolerability of a modified LD regimen, and once the maximum tolerated dose (MTD) is determined, a cohort expansion phase to further characterize the toxicity and efficacy profile and determine the recommended phase 2 dose (RP2D). The study will enroll approximately 18-24 patients in the dose escalation stage (Part 1), and approximately 20 further patients at cohort expansion (Part 2). There will be four dose escalation cohorts, in two study arms. There are two dosing cohorts in each study arm. Patients in Arm 1 will receive the ZUMA-1 chemotherapy LD regimen with or without TLI, and in Arm 2, an intermediate dose of Cy with a fixed dose of Flu, with or without TLI, will be given.

The cohorts in Arm 1 will enroll concurrently, and enrollment into Arm 2 will begin after Arm 1 has enrolled all patients and data review by the Trial Steering Committee (TSC).

For accrual into Cohort 2, Arm 1, there will be a 15-day staggered enrollment for the first 2 patients. Staggered enrollment with another 15-day delay may be considered for enrollment into Cohorts 3 and 4, Arm 2, after review by the TSC. Following completion of accrual to Arm 1, a 30 day dose-limiting toxicity (DLT) window will be observed, prior to review by the TSC and commencement of enrollment into Arm 2.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of informed consent
2. Life expectancy ≥ 12 weeks
3. Biopsy-proven and histologically confirmed R/R large B cell lymphoma, including R/R DLBCL, transformation from FL, and R/R PMBCL.
4. Radiographically documented measurable disease as per Lugano response criteria (i.e. LDi > 1.5 cm that is FDG avid).
5. At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic cancer therapy at the time the subject provides consent
6. Eligible for standard of care CAR T cell therapy, specifically, relapsed or refractory large B cell lymphoma after two or more lines of systemic therapy, and subjects must have received adequate first-line therapy including at a minimum:

   * Anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20 negative, and
   * An anthracycline containing chemotherapy regimen
7. Patient does not have active CNS disease
8. Patient is sufficiently stable to facilitate planned CAR T-cell therapy (e.g. not rapidly progressing on temporizing therapy, no significant compromise of vital organ functions (intubation, dialysis, requiring ICU/vasopressor support)) and has good performance status
9. ECOG performance status 0 or 1 at enrollment
10. Patient has not received prior adoptive T-cell immunotherapy
11. Patient is not HIV positive
12. Patient did not receive prior allogeneic stem cell transplant
13. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function
14. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
15. Sexually active males who accept to use a condom during intercourse during treatment and for 6 months after treatment as they should not father a child in this period. A condom is required to be used also by vasectomized men (as well as during intercourse with a male partner) in order to prevent delivery of the drug via seminal fluid
16. Must have an apheresis product of non-mobilized cells accepted for manufacturing.

Exclusion Criteria:

1. Persisting disease bulk (defined as ≥10 cm) on restaging imaging following bridging therapy.
2. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years
3. History of Richter's transformation of CLL
4. History of allogeneic stem cell transplant
5. Received < 2 lines of therapy for large B cell lymphoma
6. Prior CD19 targeted therapy
7. Subject has received or undergone the following:

   o Therapeutic doses of corticosteroids (defined as >20 mg/day prednisone or equivalent) within 7 days prior to leukapheresis.

   Physiologic steroid replacement, topical, and inhaled steroids are permitted.
   * Cytotoxic chemotherapeutic agents that are not considered lymphotoxic, and intrathecal (IT) chemotherapy must be stopped ≥ 7 days prior to leukapheresis.
   * Lymphotoxic chemotherapeutic agents (eg, cyclophosphamide > 300 mg/m2, ifosfamide, bendamustine) 4 weeks prior to leukapheresis.
   * Experimental agents within 4 weeks prior to signing the ICF, unless no response or PD is documented on the experimental therapy and at least 5 half-lives have elapsed prior to leukapheresis.
   * Ibrutinib, lenalidomide and PI3K inhibitor within 5 half-lives prior to leukapheresis
   * Immunosuppressive therapies within 4 weeks prior to leukapheresis (eg, calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate, rapamycin thalidomide, immunosuppressive antibodies such as anti-tumor necrosis factor [TNF], anti-IL6, or anti- IL6R)
   * Radiation within 6 weeks of leukapheresis. Subject must have progressive disease in irradiated lesions or have additional nonirradiated, PET-positive lesions to be eligible. Radiation to a single lesion, if additional non-irradiated PET-positive lesions are present, is allowed up to 2 weeks prior to leukapheresis (discuss with sponsor).
   * Treatment with systemic immunostimulatory agents (including but not limited to interferon and IL-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, prior to the infusion of axicabtagene ciloleucel
8. Prior chimeric antigen receptor therapy or other genetically modified T-cell therapy
9. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management. Simple urinary tract infection (UTI) and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
10. Known history of infection with human immunodeficiency virus (HIV) or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). If there is a positive history of treated hepatitis B or hepatitis C, the viral load must be undetectable per quantitative polymerase chain reaction (PCR) and/or nucleic acid testing.
11. Active tuberculosis
12. Presence of any indwelling line or drain (eg, percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted
13. Subjects with detectable cerebrospinal fluid malignant cells or known CNS involvement; a history of prior treated CNS lymphoma which is not active at the time of relapse is permitted
14. History or presence of significant non-malignant CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
15. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement
16. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, or other clinically significant cardiac disease within 12 months of enrollment
17. Requirement for urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression
18. History of autoimmune disease, requiring systemic immunosuppression and/or systemic disease modifying agents within the last 2 years.
19. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis per chest computed tomography (CT) scan at screening. History of radiation pneumonitis in the radiation field (fibrosis) is allowed.
20. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment
21. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
22. History of severe immediate hypersensitivity reaction to tocilizumab or any of the agents used in this study
23. Treatment with a live, attenuated vaccine within 6 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during the course of the study
24. Women of childbearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of chemotherapy on the fetus or infant.
25. Subjects of either sex who are not willing to practice birth control from the time of consent and at least 6 months after axicabtagene ciloleucel infusion
26. In the investigators judgment, the subject is unlikely to complete all protocol- required study visits or procedures, including followup visits, or comply with the study requirements for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability of chemo rads as conditioning chemo | baseline through Day 30
  To assess the safety and tolerability of a combination chemo-radiation lymphodepletion (LD) regimen (Fludarabine (Flu)/Cyclophosphamide (Cy) + total lymphoid irradiation (TLI ) in patients receiving standard of care CAR T cell therapy for relapsed/refractory diffuse large B cell lymphoma (R/R DLBCL), by establishing the maximum tolerated doses (MTD) of standard (ZUMA-1) dose Flu/Cy + TLI, and of intermediate dose iCy/Flu +/- TLI, and the dose limiting toxicities (DLT) of standard dose Flu/Cy + TLI, and of intermediate dose iCy/Flu +/- TLI

SECONDARY OUTCOMES:
Overall response rate | baseline through day 365
  The overall response rate is the proportion of patients with either a CR or PR while on study. All patients who do not meet the criteria for objective response by the analysis data cutoff date will be considered non-responders. This will be measured by CT/PET
Complete response | baseline through day 365
  To assess the efficacy (complete response (CR) rate at 12 months) of a combination chemo-radiation LD regimen (standard dose Flu/Cy + TLI) in patients receiving CAR T cell therapy for R/R DLBCL. To assess the efficacy of an intermediate dose iCy/Flu +/- TLI LD regimen in patients receiving CAR T cell therapy for R/R DLBCL. All CR and PR responses may be reviewed by an expert(s) / independent radiologist as required by simultaneous review of patient files and radiologic images
Progression free survival | baseline through day 365
  To assess the efficacy (progression free survival (PFS) at 12 months) of a combination chemo-radiation LD regimen (standard dose Flu/Cy + TLI) in patients receiving CAR T cell therapy for R/R DLBCL. To assess the efficacy of an intermediate dose iCy/Flu +/- TLI LD regimen in patients receiving CAR T cell therapy for R/R DLBCL. Progression free survival (PFS) is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada